CLINICAL TRIAL: NCT06740383
Title: Biomarkers/Biotypes, Course of Early Psychosis and Specialty Services
Acronym: BICEPS
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: University of Chicago (Other); University of Texas Southwestern Medical Center (Other); Yale University (Other); Hartford Hospital (Other); University of Georgia (Other); Mclean Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Matcheri S. Keshavan MD, Stanley Cobb Professor of Psychiatry, Beth Israel Deaconess Medical Center
Other Study IDs: 2022P000622; R01MH127174-03 (NIH)
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders; Schizophrenia; Delusional Disorder; Bipolar 1 Disorder; Schizoaffective Disorder; Psychosis Not Otherwise Specified; Early Psychosis
Keywords: schizophrenia; bipolar disorder; schizoaffective disorder; schizophreniform; major depression; psychosis; delusional disorder; Biotypes; Biomarkers; coordinated specialty care
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Schizophrenia; Schizophrenia, Paranoid; Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — venous blood samples, buccal swab samples, and immortalized lymphocyte cultures (lymphoblastoid cell lines)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Individuals with Early Psychosis enrolled in Coordinated Specialty Care Clinics: In this naturalistic longitudinal study, we administer the B-SNIP biomarker batter to individuals with Early Psychosis (EP) in EP clinics with Coordinated Specialty Care treatment programs to characterize outcome trajectories and biotypes. EP individuals of both sexes, age 18-35 will be included after they meet study criteria and provide informed consent. Individuals with psychosis duration < 3 years will be included. Individuals in this cohort of EP are diagnosed with Schizophrenia, Schizoaffective Disorder, Schizophreniform, Bipolar I Disorder with psychotic features, Delusional Disorder, Major Depressive Disorder with psychotic features, and Psychosis Not Otherwise Specified.

SUMMARY:
The Biomarkers/Biotypes, Course of Early Psychosis and Specialty Services (BICEPS) study aims to understand the early stages of psychotic disorders like Schizophrenia, Schizoaffective Disorder, and Bipolar I Disorder. It involves gathering mental health information, brain scans (MRI), eye movement patterns (Eye-Tracking), and brain electrical waves (EEG) data from individuals who have experienced these disorders in recent years. Participants will be involved for about a year, with four visits over this period. Screening procedures, lasting approximately 3 hours, include tests for drug use, a pregnancy test for eligible women, clinical interviews about feelings and experiences, psychiatric and family history interviews, and a medical history review. Research procedures for eligible participants include DNA collection, a neuropsychological test battery, EEG, eye-tracking, and MRI. These procedures will help researchers understand brain function, genetics, and cognitive abilities related to psychotic disorders. Follow-up visits at 1-month, 6-month, and 12-month intervals involve modified clinical interviews and repeating neuropsychological tests to track changes over time. Participants may opt to provide DNA samples for genetic analysis, undergo various cognitive tests, EEG to record brain waves, eye-tracking to monitor eye movements, and MRI scans to visualize brain structure. Follow-up visits at regular intervals will help researchers track changes in symptoms and cognitive function. This study provides comprehensive insight into the onset and progression of psychotic disorders and offers valuable information for patients, families, and healthcare providers involved in managing these conditions. Our goal is to better understand whether a combination of biological markers and different types of people (BT1, BT2, BT3) can help us predict how well individuals with early psychosis respond to specialized care. We expect that those in BT3 will have the best outcomes, BT2 will have intermediate outcomes, and BT1 will have the poorest outcomes. Even though BT1 and BT2 might start with similar cognitive issues, their biology might lead to different responses to treatment. This research can help us understand which treatments work best for different people with early psychosis.

DETAILED DESCRIPTION:
This proposal seeks to characterize the early course of psychotic disorders and to identify clinical and biological predictors of outcome. The large sample (=320) required will necessitate a multi-site study. All B-SNIP sites have coordinated specialty services for early course psychosis and have harmonized study procedures for uniform data collection. Each site will recruit 1/5 of the participants; The project will be managed by an all-site steering committee meeting weekly. Boston will be the coordinating site.

The outcome of early course psychosis (EP) is heterogeneous, ranging from early full recovery to treatment resistance and functional decline from the onset of illness. The ability to predict individual level outcomes would be highly valuable for treatment planning and for tailoring the duration and intensity of psychosocial and pharmacological interventions. Clinical features related to early psychosis onset are poor predictors of remission and recovery. At the same time, the field has not yet established the clinical utility of promising findings from decades of biomarker development/neuroscience research, especially in EP patients for whom empirically guided treatment planning may have the greatest impact. For example, neurocognitive, electroencephalographic (EEG) and imaging biomarkers early in the illness may predict outcome, but used individually, their prognostic value is limited. Multivariate approaches to clinical and neurobiological features may offer better value for outcome prediction.

Toward this goal, we will leverage the biomarker (EEG, eye movement testing, and neurocognition) based categorization of a cross-diagnostic sample of psychosis (biotypes) developed, replicated and validated by our Bipolar-Schizophrenia Network for Intermediate Phenotypes (B-SNIP) consortium. We have shown that Biotype-1, characterized by impaired cognition and decreased sensorimotor responses to salient stimuli is associated with the most severe impairments in functioning. Biotype-2 have the same level of cognitive impairment as Biotype-1 but increased sensorimotor reactivity. Biotype-3 cases are relatively normal on these measures and have the least impairments. These subgroups are not synonymous with DSM diagnosis and are not captured by any individual variable. We do not know if this categorization is predictive of symptomatic and functional outcome, given the cross-sectional design of B-SNIP. We will use the B-SNIP battery with EP participants in the context of Coordinated Specialty Care (CSC) treatment programs for EP available at established B-SNIP sites. Our overall goal is to identify biomarkers/Biotypes that predict clinical and functional outcome to CSC in EP. This success could guide targeted interventions in CSC programs. For those unlikely to have a successful CSC outcome, other targeted interventions could be developed and implemented. We have active EP Clinics in the consortium; each will enter about16 patients/year, 80/year overall, providing 320 EP (schizophrenia, schizoaffective disorder, psychotic bipolar disorder and schizophreniform disorder participants with approximately 240 completer cases, assuming 25% attrition) enrolled during the first 4 years of the proposed funding period. All EP cases will be tested with B-SNIP biomarker assessments at baseline, and the clinical and cognition assessments will be repeated at 1, 6, and 12 months. We will use an adapted version of the B-SNIP biomarker battery (called ADEPT) which can be implemented in under-resourced, community settings.

SIGNIFICANCE AND BACKGROUND FOR THE STUDY Schizophrenia and related psychoses cause enormous suffering for affected individual and their families and caregivers. They have a lifetime prevalence of around 3%, and cost ~ $155 billion per year in direct healthcare and indirect societal costs in the USA [5]. Relapse and poor response to treatment contribute to a significant illness burden due to high rates of hospitalization and poor social and occupational functioning. About 20% of early course psychosis (EP) cases relapse in year 1, and about 40% by year 2 [6]. Mortality is increased four-fold in EP compared to the general population [7]. EP outcomes are highly variable [8] with multiple trajectories, i.e. episodic vs persistent, initial remission vs treatment resistance [9-11]. Given this heterogeneity, actionable outcome predictors are needed to reliably individualize care for EP [12].

ELIGIBILITY:
Inclusion Criteria:

* Males and females, all races and ethnicities
* 18-35 y/o
* Meet DSM-5 criteria for a psychotic disorder, i.e. schizophrenia, schizophreniform, schizoaffective disorder, or bipolar I disorder or major depression with psychotic features, delusional disorder or psychosis N.O.S.
* Able to read, speak, and understand English
* Able and willing to provide written informed consent, and willing to commit to the study protocol
* Illness duration from psychosis onset less than or equal to 3 years

Exclusion Criteria:

* Estimated premorbid intellectual ability &lt;70 (WRAT-4, Word Reading subtest, age-corrected standardized score)
* Neurological or medical disorder that may affect brain function (seizure disorder, traumatic brain injury with a loss of consciousness greater than or equal to 3o min, history of stroke, AIDS, etc.)
* Comorbid DSM-5 diagnosis of alcohol or substance use disorders in prior 3 months (cases with cannabis use not meeting criteria for cannabis use disorder will be allowed).

MRI-Specific Exclusion Criteria:

* Pregnant women
* Presence of ferromagnetic objects in body
* Weight or body size exceeding scanner capacity (&gt;300 lbs)
* Claustrophobia

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants are recruited from 5 different sites across the United States including Boston, Dallas, Hartford, Chicago, and Georgia. The target population for this study includes individuals who meet DSM-5 criteria for a psychotic disorder (i.e., schizophrenia, schizophreniform, schizoaffective disorder, bipolar I disorder or major depression with psychotic features, delusional disorder, or psychosis N.O.S.). Participants will be between 18 and 35 years of age, males and females, of all races and ethnicities who are experiencing early course psychosis.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment Response | From enrollment at baseline to end of study at 1 year
  >30% reduction in Positive and Negative Syndrome Scale (PANSS) score
Symptomatic Remission | From enrollment at baseline to end of study at 1 year
  Score of ≤ 3 on 8 core on the Positive and Negative Syndrome Scale (PANSS) items (P1, P2, P3, 1, N4, N6, N7, G5, and G9) for at least one month
Functional Remission | From enrollment at baseline to end of study at 1 year
  Score ≥ 7 on Global Functioning Role and Social Scales
Relapse | From enrollment at baseline to end of study at 1 year
  1) Positive and Negative Syndrome Scale (PANSS) score of ≥ 4 for a psychosis item (P1, P2, P3, and P6) and ≥ 25% increase on the total PANSS score or ≥ 10 points and 2) an increased level of care, i.e. hospitalization, ER visits, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Matcheri S. Keshavan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (6):
- United States (6):
  - Hartford Hospital, Hartford, Connecticut
  - University of Georgia, Athens, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - McLean Hospital, Belmont, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The study team includes a dedicated Instructor-level faculty, Vishal Thakkar, PhD, who is responsible for data preparation and sharing. Since the beginning of the study and during the reporting period, we have been adherent with the data sharing plan and guidelines. The study has been registered in NIH/NIMH Data Archive (NDA) (Study#: C4330). Data Submission Agreement is in place. The data will be uploaded to NDA during regular data sharing cycles.
Supporting Information: Study Protocol, ICF
Time Frame: January 1st 2023 until June 30th 2028, one year after study completion
Access Criteria: The study has been registered in NIH/NIMH Data Archive (NDA) (Study#: C4330). Data Submission Agreement is in place. The data will be uploaded to NDA during regular data sharing cycles.
URL: https://www.mapnet.online/research